CLINICAL TRIAL: NCT06087003
Title: Induction Therapy of Thymoglobulin Versus Basiliximab in the Prevention of Acute Rejection After Pediatric Kidney Transplantation
Brief Title: Pediatric Induction Therapy in Kidney Transplantation
Acronym: PINK
Status: Completed | Type: Observational
Sponsor: Gang Chen (Other)
Collaborators: Zhejiang University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Changhai Hospital (Other)
Responsible Party: Sponsor-Investigator, Gang Chen, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: PINK study
Record Dates: First submitted 2023-10-08; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Kidney Transplant Rejection; Pediatric Kidney Disease
MeSH Terms: interventions — Basiliximab; thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Basilliximab induction group: Basiliximab was administered intravenously 4 hours before kidney graft reperfusion and at day 4 after kidney transplantation. For pediatric patients weighing > 30kg, the dose of Basiliximab was 20mg, otherwise was 10mg.
  Interventions: Drug: Basiliximab Injection
- rATG induction group: Rabbit antithymoglobulin (rATG) was administered intravenously during kidney transplantation (pre-reperfusion) and 1-2 days after transplantation. The dose was about 0.5-1 mg/kg per day.
  Interventions: Drug: rabbit ATG

INTERVENTIONS:
Drug: Basiliximab Injection — As an induction treatment for kidney transplantation
  Other Names: Simulect
  Groups: Basilliximab induction group
Drug: rabbit ATG — As an induction treatment for kidney transplantation
  Other Names: Thymoglobuline
  Groups: rATG induction group

SUMMARY:
The goal of this observational study is to compare the efficacy of two most commonly used induction therapy for the prevention of acute rejection (AR) after renal transplantation in children. The main question it aims to answer is:

Is basiliximab (anti-CD25 monoclonal antibody) induction therapy effective and safe in preventing AR after kidney transplantation in children compared with anti-thymoglobulin polyclonal antibodies induction therapy?

The transplant and follow-up data of participants will be retrospectively collected.

Researchers will compare the rate of AR to see if basiliximab (anti-CD25 monoclonal antibody) induction therapy is a better option for certain pediatric kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Receiving the kidney graft from a deceased donor
* Basiliximab or rATG induction therapy was used in perioperative period

Exclusion Criteria:

* Recipients with pre-transplant calculated panel reactive antibodies (cPRA) >10%
* Recipients of combined liver, pancreas or heart transplantation
* No induction or other induction therapy was used in perioperative period
* Recieving the kidney graft from a living donor

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The cohort will be selected from five centers with the highest number of pediatric kidney transplant cases in China, including Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Changhai Hospital Affiliated to Naval Medical University, the First Affiliated Hospital of Zhengzhou University, the First Affiliated Hospital of Zhejiang University and the First Affiliated Hospital of Sun Yat-sen University.
Sampling Method: Non-Probability Sample
Enrollment: 958 (Actual)
Dates: Start 2013-03-03 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Acute rejection (AR) | From baseline, kidney transplantation to data collection completion (June 30, 2023)
  The clinical diagnosis of AR is based on a significant increase in serum creatinine and the exclusion of other causes. The diagnosis of biopsy-confirmed AR is based on relevant histological changes.

SECONDARY OUTCOMES:
Cytomegalovirus (CMV) viremia | From baseline, kidney transplantation to data collection completion (June 30, 2023)
  The serum CMV is greater than 500 copies/ml
Pneumonia | From baseline, kidney transplantation to data collection completion (June 30, 2023)
  Any pneumonia that showed the presence of lesion and required hospitalization
Renal graft survival | From baseline, kidney transplantation to data collection completion (June 30, 2023)
  The estimated glomerular filtration rate (eGFR) of patient is >15 ml/min/1.73m2

CONTACTS AND LOCATIONS:
Overall Officials: Gang Chen, PhD, Principal Investigator — Tongji Hospital
Locations (5):
- China (5):
  - The First Affiliated Hospital of Sun Yat-sen University., Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhejiang University, Hangzhou
  - Changhai Hospital affiliated to Naval Military Medical University, Shanghai
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antunes H, Parada B, Tavares-da-Silva E, Carvalho J, Bastos C, Roseiro A, Nunes P, Figueiredo A. Pediatric Renal Transplantation: Evaluation of Long-Term Outcomes and Comparison to Adult Population. Transplant Proc. 2018 Jun;50(5):1264-1271. doi: 10.1016/j.transproceed.2018.02.089. PMID 29880345
- [Background] Martinez-Mier G, Enriquez-De Los Santos H, Mendez-Lopez MT, Avila-Pardo SF, Budar-Fernandez LF, Gonzalez-Velazquez F. Rejection is a strong graft survival predictor in live donor pediatric renal transplantation using cyclosporine, mycophenolate mofetil, and steroids: 5-year outcomes in a single Mexican center. Transplant Proc. 2013 May;45(4):1442-4. doi: 10.1016/j.transproceed.2013.02.044. PMID 23726592
- [Background] Crowson CN, Reed RD, Shelton BA, MacLennan PA, Locke JE. Lymphocyte-depleting induction therapy lowers the risk of acute rejection in African American pediatric kidney transplant recipients. Pediatr Transplant. 2017 Feb;21(1). doi: 10.1111/petr.12823. Epub 2016 Oct 3. PMID 27699934
- [Background] Barton KT, Halani K, Galbiati S, Dandamudi R, Hmiel SP, Dharnidharka VR; NAPRTCS investigators. Late first acute rejection in pediatric kidney transplantation: A North American Pediatric Renal Trials and Collaborative Studies special study. Pediatr Transplant. 2021 Aug;25(5):e13953. doi: 10.1111/petr.13953. Epub 2020 Dec 22. PMID 33350558
- [Background] Riad S, Jackson S, Chinnakotla S, Verghese P. Primary pediatric deceased-donor kidney transplant recipients outcomes by immunosuppression induction received in the United States. Pediatr Transplant. 2021 Aug;25(5):e13928. doi: 10.1111/petr.13928. Epub 2020 Dec 12. PMID 33314638
- [Background] Mincham CM, Wong G, Teixeira-Pinto A, Kennedy S, Alexander S, Larkins N, Lim WH. Induction Therapy, Rejection, and Graft Outcomes in Pediatric and Adolescent Kidney Transplant Recipients. Transplantation. 2017 Sep;101(9):2146-2151. doi: 10.1097/TP.0000000000001577. PMID 28832451
- [Background] Aw MM, Taylor RM, Verma A, Parke A, Baker AJ, Hadzic D, Muiesan P, Rela M, Heaton ND, Mieli-Vergani G, Dhawan A. Basiliximab (Simulect) for the treatment of steroid-resistant rejection in pediatric liver transpland recipients: a preliminary experience. Transplantation. 2003 Mar 27;75(6):796-9. doi: 10.1097/01.TP.0000054682.53834.EA. PMID 12660504
- [Background] Goh HK, Lye WC. Biopsy-proven resolution of steroid-resistant acute rejection with basiliximab therapy in a renal allograft recipient. Transplant Proc. 2001 Nov-Dec;33(7-8):3213-4. doi: 10.1016/s0041-1345(01)02368-5. No abstract available. PMID 11750379